CLINICAL TRIAL: NCT07148700
Title: Which Tools Better Predict Fall Risk in Parkinson's Disease: A Comparative Study of Objective, Self-Reported, and Functional Balance Assessment
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayça Arslantürk Yıldırım, Research Assistant, Bezmialem Vakif University
Other Study IDs: E-54022451-050.04-19466
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: PARKINSON DISEASE (Disorder); Parkinson; Parkinson s Disease; Parkinson Disease; Parkinson Disease (PD)
Keywords: Balance assessment; Functional test; Parkinson disease; Postural stability; Risk of falls
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson Disease Group: Participants diagnosed with Parkinson Disease by a neurologist

SUMMARY:
Introduction: Falls are common in Parkinson's disease (PD), affecting 30-90% of patients annually, with more than half experiencing recurrent falls. Identifying balance assessment tools that are both practical and predictive of fall risk is therefore essential. This study aimed to investigate the relationship between fall frequency and three balance assessment tools: the Biodex Balance System (objective), the Falls Efficacy Scale-International (FES-I) (self-reported), and the Mini-Balance Evaluation Systems Test (Mini-BESTest) (functional).

Methods: Patients with PD at Hoehn and Yahr stages 1-3 will be included in the study. Fall data will be collected using a fall diary, while objective balance will be assessed with the Biodex Balance System, functional performance will be evaluated with the Mini-BESTest, and self-reported balance confidence will be measured with the FES-I.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by bradykinesia, rigidity, tremor, and postural instability, resulting from damage to dopaminergic neurons in the substantia nigra. As symptom severity increases and the disease progresses, postural control deteriorates, and falls become more frequent. PD has an incidence of 13.43 per 100,000 individuals, and the number of people affected is expected to reach nine million by 2030. It has been reported that 30% to 90% of patients with PD experience at least one fall per year, with more than half of these patients experiencing recurrent falls. The etiology of falls in PD is multifactorial: age-related factors, disease-specific mechanisms, individual characteristics, and treatment-related issues all contribute to variations in fall risk among patients.

Falls in individuals with PD are associated with severe complications, including hospitalization, fear of falling, impairments in body structure and function, activity limitations, increased dependence in activities of daily living, social restrictions, and diminished quality of life. Preventing falls in PD, a problem with significant consequences and multiple risk factors, has been shown to reduce morbidity, mortality, and healthcare costs.

The fundamental strategy for preventing falls involves accurately identifying individuals at risk and initiating appropriate interventions early. Although the etiology of falls in PD appears complex, the literature suggests that balance impairments are the primary cause and that interventions should focus on improving balance. Therefore, it is crucial to identify tools that can effectively detect balance deficits. Determining the ideal balance assessment method for clinical practice requires consideration of test sensitivity, simplicity and feasibility, minimal equipment and cost requirements, ease of patient comprehension, and time efficiency. In addition, the ability of an assessment tool to accurately predict falls is a crucial criterion when selecting the most appropriate test.

Several assessments exist to assess fall risk and balance deficits in PD, including objective measures such as the Biodex Balance System, self-reported tools like the Falls Efficacy Scale-International (FES-I) and Morse Fall Scale, and functional balance tests such as the Mini-Balance Evaluation Systems Test (Mini-BESTest), Timed Up and Go Test, and Berg Balance Scale. Each of these tools has distinct advantages and disadvantages. For example, devices like the Biodex Balance System provide objective and sensitive data, but they may not reflect balance abilities during functional positions and activities of daily living, limiting their validity. Additionally, these devices require specialized equipment and can be costly.

Self-reported scales such as the FES-I are valuable as they assess an individual's perceived balance confidence during activities of daily living, including eating, personal hygiene, dressing, and transfers. However, because these assessments rely on individuals recalling their fear of falling during specific activities, responses may be influenced by memory bias or inaccurate self-perception.

Functional tests like the Mini-BESTest have the advantage of assessing task-based performance across multiple dimensions of postural control (e.g., static/dynamic balance, sensory integration, anticipatory and reactive postural adjustments) and can guide individualized treatment strategies. Nevertheless, factors such as patient motivation during testing and misunderstanding of test instructions can influence results. Functional balance tests are also time-consuming due to their multi-step structure.

Although the validity and reliability of many of these assessment tools have been established, there is insufficient evidence to determine which method best reflects actual fall risk and frequency in daily life. Furthermore, no studies have compared the predictive ability of objective, self-reported, and functional tests for future falls in patients with PD. The aim of this study is to investigate the relationship between fall frequency and three different tools for balance assessment: the Biodex Balance System, which provides objective measurements; the FES-I, which relies on self-reported data; and the Mini-BESTest, which evaluates functional balance performance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years old
* Receiving stable dopaminergic treatment
* No other neurological disorders besides PD
* A Standardized Mini-Mental State Examination (MMSE) score >24
* Hoehn and Yahr stage between 1-3
* Voluntarily agreed to participate in the study after receiving detailed information

Exclusion Criteria:

Presence of visual, hearing impairments, cardiovascular or pulmonary diseases that could affect study outcomes

* Having mental or physical impairments severe enough to hinder communication
* Clinically unstable condition within the past month
* Participation in a rehabilitation program within the last six months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with PD by a neurologist and meeting the following criteria
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Fall Diary | At baseline (immediately after informed consent)
  A "Fall Diary" is used as a retrospective interview tool to collect information on falls that have occurred during the previous six months. Participants are asked to recall and report the number of falls within this period, along with details regarding the activity being performed at the time of the fall, the environmental context, balance strategies attempted during the fall, the method of recovery, the occurrence of any complications, and whether medical assistance or hospitalization is required. To enhance the accuracy and completeness of the retrospective fall reports, caregivers are also consulted to corroborate and supplement the participants' accounts.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale-III (UPDRS-III) | At baseline (immediately after informed consent)
  The UPDRS, developed by the Movement Disorder Society, is used as a comprehensive and widely accepted clinical tool for evaluating PD. The third part of the scale, the Motor Examination section, is utilized in this study. This section evaluates motor symptoms including speech, facial expression, rigidity, finger tapping, hand movements, pronation-supination, toe tapping, leg agility, rising from a chair, gait, freezing of gait, postural stability, posture, trunk bradykinesia, postural tremor, kinetic tremor, resting tremor amplitude, tremor constancy, and impact of dyskinesia. It consists of 18 items scored between 0 and 4, with higher scores indicating greater symptom severity. The validity and reliability of the Turkish version have previously been established.
Mini-Balance Evaluation Systems Test (Mini-BESTest) | At baseline (immediately after informed consent)
  The Mini-BESTest is used as a valid and reliable clinical tool for functionally evaluating balance in individuals with PD. The test consists of 14 items across four subdomains: anticipatory postural adjustments (APA), reactive postural control (RPC), sensory orientation (SO), and dynamic gait (DG). It is scored out of 28 points and takes approximately 10-15 minutes to complete. Higher scores indicate better balance performance. Strong inter-rater and test-retest reliability as well as high concurrent validity compared with the original BESTest are being demonstrated in previous studies.
Biodex Balance System (BBS)-Postural Stability Test (PST) | At baseline (immediately after informed consent)
  This test is used to assess participants' ability to maintain their center of balance on a static platform by measuring their deviations from the center. The overall stability index (OSI) reflects total variability, the anterior-posterior index (APSI) represents sagittal plane variability, and the medial-lateral index (MLSI) indicates frontal plane deviations. Higher scores indicate greater impairment in postural stability. The test is conducted over three trials, each lasting 30 seconds, with a 15-second rest between trials.
Biodex Balance System (BBS)-Fall Risk Index (FRI) Test | At baseline (immediately after informed consent)
  The FRI test involves a progressive protocol transitioning from a stable to an unstable surface and measures deviations from the center to calculate a fall risk index. In this study, the platform setting is fixed at level 12-1 for all participants.
Falls Efficacy Scale-International (FES-I) | At baseline (immediately after informed consent)
  The FES-I is used to assess participants' concerns about falling during physical and social activities. The Turkish version of the scale has been validated. It consists of 16 items, each rated on a 4-point Likert scale ("not at all concerned," "somewhat concerned," "fairly concerned," "very concerned"), with total scores ranging from 16 to 64. Higher scores reflect greater fear of falling. The FES-I is reported to demonstrate excellent reliability in individuals with PD, both in the "on" (ICC = 0.94) and "off" (ICC = 0.91) drug phases.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyup, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share IPD: Yes. Individual participant data (IPD) that underlie the results reported in the article (after de-identification) will be shared. This will include baseline characteristics data, and outcome measures.
  What data will be shared: De-identified individual participant data related to primary and secondary outcomes.
  When data will be available: Beginning 6 months after publication of the main results and ending 5 years after publication.
  How data will be shared: Data will be made available upon reasonable request to the corresponding author, after approval of a research proposal and signing of a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months after publication of the main results and ending 5 years after publication.
Access Criteria: Data will be made available upon reasonable request to the corresponding author, after approval of a research proposal and signing of a data access agreement.

REFERENCES:
- [Background] Winser SJ, Kannan P, Bello UM, Whitney SL. Measures of balance and falls risk prediction in people with Parkinson's disease: a systematic review of psychometric properties. Clin Rehabil. 2019 Dec;33(12):1949-1962. doi: 10.1177/0269215519877498. Epub 2019 Oct 1. PMID 31571503
- [Background] Meekes WM, Korevaar JC, Leemrijse CJ, van de Goor IA. Practical and validated tool to assess falls risk in the primary care setting: a systematic review. BMJ Open. 2021 Sep 29;11(9):e045431. doi: 10.1136/bmjopen-2020-045431. PMID 34588228
- [Background] Lopes LKR, Scianni AA, Lima LO, de Carvalho Lana R, Rodrigues-De-Paula F. The Mini-BESTest is an independent predictor of falls in Parkinson Disease. Braz J Phys Ther. 2020 Sep-Oct;24(5):433-440. doi: 10.1016/j.bjpt.2019.07.006. Epub 2019 Jul 25. PMID 31377123
- [Background] Schlenstedt C, Brombacher S, Hartwigsen G, Weisser B, Moller B, Deuschl G. Comparison of the Fullerton Advanced Balance Scale, Mini-BESTest, and Berg Balance Scale to Predict Falls in Parkinson Disease. Phys Ther. 2016 Apr;96(4):494-501. doi: 10.2522/ptj.20150249. Epub 2015 Sep 17. PMID 26381806
- [Background] Liu WY, Tung TH, Zhang C, Shi L. Systematic review for the prevention and management of falls and fear of falling in patients with Parkinson's disease. Brain Behav. 2022 Aug;12(8):e2690. doi: 10.1002/brb3.2690. Epub 2022 Jul 14. PMID 35837986
- [Background] Camicioli R, Morris ME, Pieruccini-Faria F, Montero-Odasso M, Son S, Buzaglo D, Hausdorff JM, Nieuwboer A. Prevention of Falls in Parkinson's Disease: Guidelines and Gaps. Mov Disord Clin Pract. 2023 Sep 2;10(10):1459-1469. doi: 10.1002/mdc3.13860. eCollection 2023 Oct. PMID 37868930
- [Background] Schrag A, Choudhury M, Kaski D, Gallagher DA. Why do patients with Parkinson's disease fall? A cross-sectional analysis of possible causes of falls. NPJ Parkinsons Dis. 2015 Jun 11;1:15011. doi: 10.1038/npjparkd.2015.11. PMID 28409181
- [Background] Kerr GK, Worringham CJ, Cole MH, Lacherez PF, Wood JM, Silburn PA. Predictors of future falls in Parkinson disease. Neurology. 2010 Jul 13;75(2):116-24. doi: 10.1212/WNL.0b013e3181e7b688. Epub 2010 Jun 23. PMID 20574039
- [Background] Ou Z, Pan J, Tang S, Duan D, Yu D, Nong H, Wang Z. Global Trends in the Incidence, Prevalence, and Years Lived With Disability of Parkinson's Disease in 204 Countries/Territories From 1990 to 2019. Front Public Health. 2021 Dec 7;9:776847. doi: 10.3389/fpubh.2021.776847. eCollection 2021. PMID 34950630
- [Background] Dorsey ER, Bloem BR. The Parkinson Pandemic-A Call to Action. JAMA Neurol. 2018 Jan 1;75(1):9-10. doi: 10.1001/jamaneurol.2017.3299. No abstract available. PMID 29131880